CLINICAL TRIAL: NCT02286934
Title: A Clinical Trial to Investigate the Influence of Cytochrome P450 2D6 Polymorphism on the Pharmacokinetic/Pharmacodynamics Characteristics of Carvedilol in Healthy Korean Volunteers
Brief Title: Cytochrome P450 2D6 Genotype on the Clinical Effect of Carvedilol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Institute of Food and Drug Safety Evaluation, Korea (Unknown)
Responsible Party: Principal Investigator, Jae Yong Chung, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYP-CVDL-01
Record Dates: First submitted 2014-09-05; First posted 2014-11-10 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Carvedilol; CYP2D6; Isoproterenol Sensitivity Test
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carvedilol (Experimental): * Day 1 to 3 : Carvedilol 12.5 mg qd
  * Day 4 to 8 : Carvedilol 25 mg qd
  * Day 9 to 11 : Carvedilol 12.5 mg qd
  Isoproterenol Sensitivity Test
  * Day 0, 1.5h post-dose Injection of isoproterenol 4 times (0.25, 0.5, 1, 2 ug/mL), time interval of 10 minutes.
  * Day 1, 8, 1.5h post-dose Injection of isoproterenol 4 times (5, 10, 20, 40 ug/mL), time interval of 10 minutes.
  Measure change of heart rates after 1, 2, 3 minutes post injection of isoproterenol.
  Interventions: Drug: Carvedilol; Other: Isoproterenol Sensitivity Test

INTERVENTIONS:
Drug: Carvedilol — * Day 1 to 3 : Carvedilol 12.5 mg qd
  * Day 4 to 8 : Carvedilol 25 mg qd
  * Day 9 to 11 : Carvedilol 12.5 mg qd
Other: Isoproterenol Sensitivity Test — Day 0, 1, 8 : Isoproterenol Sensitivity Test

SUMMARY:
A Clinical Study to Evaluate the Effect of Cytochrome P450 2D6 polymorphism on Pharmacokinetics/Pharmacodynamics After Multiple Administration of Carvedilol

DETAILED DESCRIPTION:
This study has an open-label, one-sequence, multiple drug administration design. The purpose of this study is as follows;

To evaluate the change of the result of Isoproterenol Sensitivity Test according to Cytochrome P450 2D6 genotype after the multiple administration of carvedilol

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects aged 20 - 45 years
* A body mass index (BMI) in the range 18.0 kg/m2 (inclusive) - 27.0 kg/m2 (inclusive).
* Sufficient ability to understand the nature of the study and any hazards of participating in it. Provide written informed consent after being fully. informed about the study procedures.

Exclusion Criteria:

* Presence or history of hypersensitivity or allergic reactions to drugs including investigational product (Carvedilol, Isoproterenol).
* Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AUC (area under the plasma concentration-time curve) of carvedilol | predose and 0.25, 0.5, 1, 2, 3, 4, 6, 12, 24h postdose
Cmax (Maximum plasma concentration) of carvedilol | predose and 0.25, 0.5, 1, 2, 3, 4, 6, 12, 24h postdose

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, MD, PhD, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University Bundang Hospital, Seongnam, Kore
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyounggi, South Korea

REFERENCES:
- [Derived] Jung E, Ryu S, Park Z, Lee JG, Yi JY, Seo DW, Lee J, Jeong HS, Kim JM, Oh WY. Influence of CYP2D6 Polymorphism on the Pharmacokinetic/Pharmacodynamic Characteristics of Carvedilol in Healthy Korean Volunteers. J Korean Med Sci. 2018 May 23;33(27):e182. doi: 10.3346/jkms.2018.33.e182. eCollection 2018 Jul 2. PMID 29962926